CLINICAL TRIAL: NCT02748200
Title: Muscle Invasive Bladder Cancer: External Beam Radiotherapy as an Alternative for Cystectomy
Brief Title: External Beam Radiotherapy for Muscle Invasive Bladder Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/0169
Record Dates: First submitted 2015-03-18; First posted 2016-04-22 (Estimated); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Toxicity

STUDY DESIGN:
Intervention Model Description: All patients receive pelvic EBRT to the lymph nodes located along the common, internal, and external iliac artery; obturator fossa; and presacral nodes.
Oversight: Data Monitoring Committee: No

ARMS (3):
- external beam radiotherapy: Dose level 1 (Experimental): 57.6 Gray (Gy) (20 x 2.88 Gy, 5 fractions/week, 4 weeks)
  Interventions: Radiation: external beam radiotherapy (EBRT)
- external beam radiotherapy: dose level 2 (Experimental): 60 Gy (20 x 3.00 Gy, 5 fractions/week, 4 weeks)
  Interventions: Radiation: external beam radiotherapy (EBRT)
- external beam radiotherapy: dose level 3 (Experimental): 62.4 Gy (20 x 3.12Gy, 5 fractions/week, 4 weeks)
  Interventions: Radiation: external beam radiotherapy (EBRT)

INTERVENTIONS:
Radiation: external beam radiotherapy (EBRT) — EBRT: 3 dose escalation levels

SUMMARY:
In this phase 1 trial, the investigators will prospectively evaluate 3 different external beam radiotherapy (EBRT) schedules. In every schedule, the whole bladder will be treated to 40 Gray (Gy) in 20 fractions, 5 fractions/week, 4 weeks in total. Based on the summation of abnormalities seen on pre- (initial tumor region) and post transurethral resection zone of fibrosis Diffusion weighted-magnetic resonance imaging (MRI) images the tumor region is delineated and defined as a gross tumor volume (GTV). The GTV will be treated using a simultaneous integrated boost (SIB): without extending the 4-weeks treatment period, 3 different dose levels will be implemented in order to increase the biological equivalent dose (BED), as muscle invasive bladder cancer has been shown to be dose-sensitive.

DETAILED DESCRIPTION:
3 different dose levels will be implemented in order to increase the biological equivalent dose (BED), as muscle invasive bladder cancer has been shown to be dose-sensitive.

* Level 1: 57.6 Gray (Gy) (20 x 2.88 Gy, 5 fractions/week, 4 weeks); BED: 61 Gy.
* Level 2: 60 Gy (20 x 3.00 Gy, 5 fractions/week, 4 weeks); BED: 64 Gy
* Level 3: 62.4 Gy (20 x 3.12Gy, 5 fractions/week, 4 weeks); BED: 67 Gy. Fiducials will be implanted at the edges of the postoperative bed during the second transurethral resection of the bladder to improve visualization of the gross tumor volume (GTV) during external beam radiotherapy (EBRT) and consequently improve treatment delivery accuracy. In order to further improve the treatment accuracy, 5 planning Computed Tomographies and plans, with different bladder fillings will be made upfront in our study. During treatment the plan corresponding best with bladder filling at time of EBRT will be selected and delivered.

ELIGIBILITY:
Inclusion Criteria:

* histological proven diagnosis of muscle invasive bladder cancer
* stage <T3b tumours with pathological lymph nodes after extended pelvic lymph node dissection
* World Health Organisation performance state 0-2
* signed informed consent

Exclusion Criteria:

* contra-indication for Diffusion-Weighted-Magnetic resonance imaging

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Radiation Therapy Oncology Group toxicity scale | 3 months after radiotherapy

SECONDARY OUTCOMES:
Number of participants free from local relapse assessed on cystoscopy and Magnetic Resonance Imaging | 12 months after radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Fonteyne, MD; PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided